CLINICAL TRIAL: NCT07273071
Title: Individualized Multiplex Pathophysiological Treatment of Severe Acute Infections (IMPACT): A Randomized, Open-Label Clinical Trial to Assess Whether an Individualized Treatment Strategy Aimed at Preventing Organ Dysfunction Can Reduce Mortality and Decrease Hospital Length of Stay in Patients With Severe Acute Infections
Brief Title: Individualized Multiplex Pathophysiological Treatment of Severe Acute Infections
Acronym: IMPACT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Theis S. Itenov (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Sponsor-Investigator, Theis S. Itenov, Clinical Associate Professor and Specialist Physician, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-522215-42-00; 2025-522215-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Acute Infection; Severe Infection
Keywords: Sepsis; Acute Infection; Severe Infection; Individualized Treatment; Treatment Bundle; CPAP; Ketone Ester; Acetylcysteine; Iron; Hydrocortisone
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Masking Description: The person performing the EQ-5D-5L questionnaire is masked to treatment allocation. The DSMB is masked to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Treatment Strategy (Experimental)
  Interventions: Combination Product: Individualized Treatment Strategy
- Standard-of-care (No Intervention)

INTERVENTIONS:
Combination Product: Individualized Treatment Strategy — An individualized treatment strategy, where the participant receives up to five of the following: continuous positive airway pressure (CPAP), ketone ester, N-acetylcysteine, iron infusion, hydrocortisone. Each participant's bundle is defined by results from an extended clinical examination.
  Arms: Individualized Treatment Strategy

SUMMARY:
The goal of the IMPACT trial is to determine whether an individualized treatment strategy, initiated at admission to the Emergency Department, can reduce hospitalizations and improve survival among patients with sepsis. To address this question, we will enroll 300 participants in a randomized controlled trial.

All participants will undergo an extended clinical assessment. Those randomized to the individualized treatment arm may receive up to five targeted interventions, depending on the findings of this assessment.

The targeted interventions are:

1. Continuous positive airway pressure (CPAP) to support breathing and help prevent respiratory problems in participants who show signs of breathing difficulties on ultrasound.
2. Ketone ester, a nutritional supplement, to help support heart function in participants who show signs of heart strain on ultrasound.
3. N-acetylcysteine, an antioxidant treatment, to help protect the liver in participants with early signs of liver stress.
4. Intravenous iron to help prevent or treat anemia in participants who show signs of low iron levels.
5. Hydrocortisone, a steroid, to help stabilize the immune system in participants with signs of immune overactivation.

Participants randomized to the control group will receive standard-of-care according to local clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Suspected acute infection within 72 hours of admission, defined as (1) having samples collected for bacterial isolation and/or (2) being initiated on antibiotic therapy
3. Documented clinical suspicion of infection
4. Admitted to the hospital with an expected duration greater than 24 hours
5. Sequential organ failure assessment (SOFA) score ≥2

Exclusion Criteria:

1. Informed consent following inclusion expected to be unobtainable
2. Inability to read and understand Danish to a degree that allows valid informed consent and completion of trial assessments
3. Pregnant or breastfeeding patients
4. Involuntary admission under the psychiatric law
5. Admitted to hospital or undergone surgery during the 14 days prior to admission
6. Expected initiation of palliative care within 48 hours of randomization
7. Previous randomization into the current trial
8. Admitted to ICU or expected transfer to ICU within 2 hours
9. Previous severe anaphylaxis
10. Any other condition deemed by the investigator to compromise patient safety or trial integrity (e.g., severe coagulopathy, uncontrolled bleeding, diabetic ketoacidosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital at 14 days post-randomization (DAOH-14) | Assessed 14 days post-randomization

SECONDARY OUTCOMES:
Number of participants with one or more serious adverse event within 14 days of randomization | Assessed 14 days post-randomization
Days alive and out of hospital at 30 days post-randomization | Assessed 30 days post-randomization
All-cause mortality at 14, 30 and 180 days after inclusion | Assessed at 14, 30 and 180 days post-randomization
ICU admission within 14 and 30 days of randomization | Assessed at 14 and 30 days post-randomization
Hospital length of stay within 14 and 30 days of randomization | Assessed at 14 and 30 days post-randomization
Health related quality-of-life at 180 days post-randomization (EQ-5D-5L) | Assessed 180 days post-randomization
Duration of antibiotic therapy within 14 and 30 days of randomization | Assessed at 14 and 30 days post-randomization
Escalation of antibiotic therapy within 14 and 30 days of randomization | Assessed at 14 and 30 days post-randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, Copenhagen University Hospital - Bispebjerg and Frederiksberg, Copenhagen, Denmark